CLINICAL TRIAL: NCT07227896
Title: A Global Real-World Evidence Study on the Effectiveness and Safety/Tolerability of Foslevodopa/Foscarbidopa in Patients Earlier Within Advanced Parkinson's Disease
Brief Title: Real-World Study of Foslevodopa/Foscarbidopa to Assess Quality of Life Outcomes in Adult Participants Earlier Within Advanced Parkinson Disease
Acronym: PUCCINI
Status: Not yet recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-758
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Foslevodopa/Foscarbidopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foslevodopa/Foscarbidopa: Participants will receive Foslevodopa/Foscarbidopa as prescribed by their physician according to local label.

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how effective Foslevodopa/Foscarbidopa is in treating adult participants earlier within advanced Parkinson disease under routine clinical practice.

Foslevodopa/Foscarbidopa is an approved drug for the treatment of Parkinson's Disease. Approximately 100 adult participants who are prescribed Foslevodopa/Foscarbidopa by their doctors will be enrolled across approximately 40 sites across the world.

Participants will receive Foslevodopa/Foscarbidopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 6 months.

There are no additional examinations due to the study but the participants and caregivers will need to fill several questionnaires to generate data on their motor function and well-being

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for Foslevodopa/Foscarbidopa (LDp/CDp) therapy in accordance with approved local label in the participating country and local reimbursement regulations, if applicable
* A diagnosis of levodopa-responsive idiopathic Parkinson's Disease (PD)
* Adult male or female between 18 and 80 years of age
* Disease duration (time since diagnosis) <10 years
* Time since motor fluctuations ≤3 years
* H&Y Stage <3 in best "on"
* "off" time of 2.5-6 hours per day
* Naïve to LDp/CDp
* Treatment has been optimized with oral/transdermal PD medication in the opinion of the Investigator
* Decision to treat with LDp/CDp made by the clinician prior to any decision to approach the participant to participate in the study
* Willing and able to comply with procedures required during this study, specifically with entering data and filling questionnaires in an electronic device (tablet).
* Prior to any study-related procedures being performed, the participant or Legal Authorized Representative (LAR) must voluntarily sign an Authorization for Use/Disclosure of Data (AUDD)/Informed Consent Form (ICF) according to national regulations once the study has been explained and the participant has the opportunity to have any questions answered

Exclusion Criteria:

* History of any condition included in the contraindications section of the approved local Foslevodopa/Foscarbidopa (LDp/CDp) label in the participating country
* History of treatment with any Device-Aided Therapy (DAT), such as Deep Brain Stimulation (DBS), Continuous Subcutaneous Apomorphine Infusion (CSAI), Levodopa/Carbidopa Intestinal Gel (LCIG)/ Carbidopa/Levodopa Enteral Suspension (CLES), Levodopa/Entacapone/Carbidopa Intestinal Gel (LECIG)
* Mini-Mental State Examination (MMSE) score <24
* Participation in a concurrent investigational or observational clinical trial
* Lack of motivation/insufficient language skills to complete the study questionnaires
* History of significant skin conditions or disorders (e.g., psoriasis, atopic dermatitis). In case of temporary affections like recent sunburn or open wounds, or in case of permanent affections like acne, scar tissue, tattoo, branding, or colorations, the participant should not be included if the Investigator considers these as interfering with infusion of study drug or study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with earlier within advanced Parkinson disease receiving Foslevodopa/Foscarbidopa treatment in accordance with the local label requirements in the participating country.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in OFF Time (hours) as measured by modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) IV | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD)

SECONDARY OUTCOMES:
Change From Baseline in Dyskinesia presence as measured by modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) IV | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). (The numeric score for each question is between 0-4; 0=Normal, 4=Severe)
Change From Baseline in Dyskinesia duration (absolute hours) as measured by modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) IV | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD).
Change From Baseline in Motor complications as measured by modified Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) IV | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). (The numeric score for each question is between 0-4; 0=Normal, 4=Severe)
Change From Baseline in Disease-specific Quality of Life (QoL) as measured by the Parkinson's Disease Questionnaire-39 Items (PDQ-39) Summary Index | Up to approximately 6 months
  The Parkinson's Disease Questionnaire (PDQ-39) is a disease-specific instrument designed to measure aspects of health that are relevant to participants with Parkinson's Disease (PD), and which may not be included in general health status questionnaires. Each item is scored on the following 5-point scale: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always (or cannot do at all, if applicable).
Change From Baseline in Generic Quality of Life (QoL) as measured by the EuroQol 5-Dimension Questionnaire (EQ-5D-5L) | Up to approximately 6 months
  The EuroQol 5-dimension questionnaire (EQ-5D-5L) is a standardized non-disease specific instrument for describing and valuing health-related quality of life. The EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the participant's current health state. Each item is scored from 1 (best) to 5 (worst). An increase in the EQ-5D-5L score indicates a worsening.
Change From Baseline in Motor experiences of daily living as measured by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Up to approximately 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). Part II assesses the participant's motor experiences of daily living (M-EDL) with 13 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part II scores range from 0 to 52, with higher scores indicating more severe symptoms of PD. Negative changes from Baseline indicate improvement.
Change From Baseline in Disease-specific sleep disturbances as measured by the Parkinson's Disease Sleep Scale-2 (PDSS-2) Total Score | Up to approximately 6 months
  The PDSS-2 consists of 15 questions that evaluate motor and non-motor symptoms at night and upon wakening, as well as disturbed sleep grouped into 3 domains: motor symptoms at night (5 items), Parkinson's Disease (PD) symptoms at night (5 items), and disturbed sleep (5 items). The frequency is assessed for the 15 sleep problems based on a 5-point Likert-type scale (ranging from 0 [never] to 4 [very often] with the exception of Question 1 score ranging from 0 [very often] to 4 [never]).
Change From Baseline in Symptom severity measured by the Patient Global Impression of Severity (PGI-S) | Up to approximately 6 months
  The Patient Global Impression of Severity (PGI-S) is a single, patient-reported item that assesses the subject's perceived level of symptoms over the past 7 days. The measure uses a 5-point Likert rating scale with responses ranging from "no symptoms" (1) to "very severe" (5), with higher scores indicating greater severity.
Change From Baseline in Symptom severity measured by the Patient Global Impression of Change (PGI-C) | Up to approximately 6 months
  The Patient Global Impression of Change (PGI-C)is a 7-point response scale. The participant was asked by the Investigator or qualified designee to rate their change in status using the following 7-point scale: Scores range from 1 = Very much improved; to 7 = Very much worse.
Change From Baseline in Symptom severity measured by the Clinical Global Impression of Severity (CGI-S) scores | Up to approximately 6 months
  Clinical Global Impression of Severity (CGI-S) is a 7-point rating scale used to measure the that requires the clinician to assess how much the participant's illness has improved or worsened relative to the baseline state at the beginning of the intervention. Scores range from 1=normal; to 7=among the most extremely ill.
Change From Baseline in Symptom severity measured by the Clinical Global Impression of Change (CGI-C) scores | Up to approximately 6 months
  The Clinical Global Impression of Change (CGI-C) is a clinician's impression of a subject's change in status on a 7-point scale. CGI-C scores range from 1 = very much improved to 7 = very much worse.

OTHER OUTCOMES:
Change From Baseline in morning akinesia (early morning "off") as measured by by dedicated questionnaire. | Up to approximately 6 months
  Measured by dedicated questionnaire.
Change From Baseline in Activities of daily living/independence as measured by the Schwab-England Activities of Daily Living Scale (SE-ADL) | Up to approximately 6 months
  Schwab-England Activities of Daily Living Scale (SE-ADL) onsists of ten items intended to evaluate the daily life activities of a participant. The SEADL is composed of two sections: the first is a self-reported questionnaire in which participants grade their own daily life activities, such as dressing, using the toilet, resting, eating, and social activities (subjective assessment), and the second is an assessment of motor functions, such as postural balance, speaking, rigidity, and tremors, conducted by a clinician (objective assessment). It is a percentage scale divided into deciles, and the results are reported between 0% (bedridden) and 100% (healthy). Negative changes in values indicate a decline in health.
Change From Baseline in Self-efficacy as measured by the Self-efficacy for Managing Chronic Disease Scale (SEMCD) | Up to approximately 6 months
  Self-efficacy for Managing Chronic Disease Scale (SEMCD) Self-efficacy for chronic disease will be measured.
Change From Baseline in Ability to reintegrate into normal social activity after illness as measured by the Reintegration to Normal Living Scale (RNLI) Scale | Up to approximately 6 months
  Reintegration to Normal Living Scale (RNLI) Scale the reintegrate into normal social activity after illness will be measured
Change From Baseline in Treatment satisfaction, as measured by the Treatment Satisfaction Questionnaire for Medication, 9-Item Version Score (TSQM-9) | Up to approximately 6 months
  Treatment Satisfaction Questionnaire for Medication, 9-Item Version Score. an instrument to show that adherence is expected to be related with participants' satisfaction with therapy and that such satisfaction can be a function of not only the effect of the treatment, but also the services offered. Range of the domain scores range from 0 to 100 with higher scores indicating a better state or outcome (e.g., greater perceived effectiveness or satisfaction).
Change From Baseline in Stigma as measured by the Parkinson's Disease Questionnaire-39 Items (PDQ-39) Summary Index | Up to approximately 6 months
  The Parkinson's Disease Questionnaire (PDQ-39) is a disease-specific instrument designed to measure aspects of health that are relevant to participants with Parkinson's Disease (PD), and which may not be included in general health status questionnaires. Each item is scored on the following 5-point scale: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always (or cannot do at all, if applicable).
Number of Participants who used Healthcare Resource Utilization (HRU) | Up to approximately 6 months
  HRU is measured from initiation of the studied line of therapy and captures .. eg physician visits, hospital stays and engagement with other supporting therapists.
Number of Participants achieving monotherapy with Foslevodopa/Foscarbidopa (LDp/CDp) | Up to approximately 6 months
  Percentage of patients achieving monotherapy with LDp/CDp at month 3 and month 6
Questionnaire to investigate the practicalities of the infusion system | Up to approximately 6 months
  Questionnaire to investigate the practicalities of the infusion system e.g., vial consumption, frequency of infusion-site rotation, nighttime dose adjustments) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Boston Medical Center Health System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-758